CLINICAL TRIAL: NCT06711016
Title: Cerebral Perfusion and Oxygenation-oriented Multimodal Neurological Monitoring Strategy for Patients with Refractory Out-of -hospital Cardiac Arrest (OHCA)
Brief Title: Multimodal Neurological Monitoring Strategy After Receiving ECPR
Acronym: MNM-ECPR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: China-Japan Friendship Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); Second Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Feng Xu, Professor, Qilu Hospital of Shandong University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: KYLL-202409-012-1
Record Dates: First submitted 2024-11-04; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-08

CONDITIONS: Cardiac Arrest
Keywords: Multimodality Neuromonitoring; ECPR; Out-of-hospital Caridac arrest
MeSH Terms: conditions — Heart Arrest | interventions — Anticonvulsants; Equipment and Supplies

STUDY DESIGN:
Intervention Model Description: The control group: The goals of resuscitation include radial oxygen saturation between 92 and 98%, MAP ≥ 65 mmHg, Hb ≥ 7 g/dL, pH 7.35 to 7.45, and coagulation in accordance with ECMO management requirements. Routine fluid resuscitation, dehydration and intracranial pressure reduction, ECMO circulatory flow adjustment, temperature management, ventilator-supported ventilation, coronary angiography if coronary causes are suspected.
  The experimental group：The Vm will maintained between 56-85 cm/s, Vd>30cm/s，PI <1.2, the cerebral oxygen saturation (rSO2) in the brain region will maintained between 60%-70%, ONSD<5.5mm, and the pathological state will be monitored with EEG by regulating the ECMO parameters, temperature treatment, ventilation, vasoactive agent, sedative and antiepileptic drug et al. if necessary. The rest were monitored and treated with the control group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- multimodal monitoring strategy (Experimental): These include TCD to monitor cerebral blood perfusion levels, NIRS to monitor oxygen saturation levels in brain regions, ONSD to evaluate cerebral edema, and continuous quantitative EEG to monitor brain function to assess prognosis. Among them, The Vm will maintained between 56-85 cm/s, Vd>30cm/s，PI<1.2, the cerebral oxygen saturation (rSO2) in the brain region will maintained at 55%-75%, ONSD <5.5mm, and the pathological state will be monitored with EEG.
  Interventions: Other: fluid resuscitation, vasoactive drug dose,hemoglobin transfusion,sedative analgesic muscle relaxant drugs, antiepileptic drugs, etc
- control (Active Comparator): SPO2 between 92 and 98%, MAP ≥ 65 mmHg, Hb ≥ 7 g/dL, pH 7.35 to 7.45, Pco2 between 40-45 mmHg， Routine fluid resuscitation, dehydration and intracranial pressure reduction, ECMO circulatory flow adjustment, temperature management, ventilator-supported ventilation, coronary angiography if coronary causes are suspected.
  Interventions: Other: fluid resuscitation, vasoactive drug dose,hemoglobin transfusion,sedative analgesic muscle relaxant drugs, antiepileptic drugs, etc

INTERVENTIONS:
Other: fluid resuscitation, vasoactive drug dose,hemoglobin transfusion,sedative analgesic muscle relaxant drugs, antiepileptic drugs, etc — ECMO flow, IABP , ventilator support parameters, temperature management level and time
  Other Names: Device

SUMMARY:
Neurological injury remains an important cause of morbidity and mortality in patients with ECPR. At present, the results of three prospective randomized controlled studies on ECPR are inconsistent, and it is inconclusive whether ECPR can improve the neurological outcomes of patients with refractory cardiac arrest. Several study found that extracorporeal membrane oxygenation nonsurvivors can lead toacute brain injury.Further research with a systematic neurologic monitoring is necessary to define the timing of acute brain injury in patients with extracorporeal membrane oxygenation.Moreover, brain injury that occurs during extracorporeal membrane oxygenation therapy is not easy to detect in time because of the use of analgesics, sedatives, and muscle relaxants. Surprisingly, little attention has been paid to the role of cerebral perfusion and oxygenation. Moreover,the features of cerebrovascular pathophysiology and optimal management strategies are still vague.

Therefore multimodal neuromonitoring may be a valuable tool for detecting brain injury in patients with extracorporeal membrane oxygenation and providing early intervention guidance.

The aim of this study is to test whether multimodal neuromonitoring will improve 30-day survival with a favorable neurologic outcome in ECPR patients with a refractory OHCA.

ELIGIBILITY:
Inclusion Criteria:

1. Presumed or known to be 18-75 years old
2. Witnessed OHCA
3. Initially presenting with VF/VT or who have been administered an AED-shock
4. Bystander CPR
5. No flow time (time from CA to CPR) was less than 5 min
6. Fail to achieve sustained ROSC within 15 minutes

Exclusion Criteria:

1. ROSC with sustained hemodynamic recovery within 15 minutes
2. Terminal heart failure (NYHA III or IV), severe pulmonary disease (COPD Gold III or IV), oncological disease,
3. Pregnancy
4. Bilateral femoral bypass surgery
5. Pre arrest Cerebral Performance Category (CPC) score of 3 or 4
6. Multiple trauma (Injury Severity Score>15)
7. Estimated that cannulation will start 90 minutes after the initial arrest.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 654 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2028-05-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
30-day survival rate with favorable neurological status | 30 days
  Cerebral Performance Category (CPC) score will be performed to evaluate the neurological status. A CPC score of 1 or 2 indicates a favorable neurological status.

SECONDARY OUTCOMES:
Survival with favorable neurological status at 3, 6 months | 3 months, 6 months
  Does multimodal neurological monitoring Strategy improve the neurological outcome at 3 months, 6 months.
  A Cerebral Performance Category (CPC) score of 1 or 2 indicates a favorable neurological status.
Time to return of circulation | Within 1 year
  What is the time to return of circulation
Duration of mechanical ventilation | 1 year
  Is there a difference in the duration of mechanical ventilation between treatment groups
Length of stay at the ICU | 1 year
  Is there a difference in length of stay at the ICU between the treatment groups
Length of stay at the hospital | 1 year
  Is there a difference in length of stay at the hospital between the treatment groups
Duration of hypothermia | 1 year
  Is there a difference in duration of hypothermia between the treatment groups
Difference in NSE, S100 B level between treatment groups | 3 days
  Is there a difference in nerve damage Markers such as (1) NSE, (2) S100B at ROSC 24h, 48h, 72h between the treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Yuguo Chen, MD. PhD, Study Chair — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No